CLINICAL TRIAL: NCT05059028
Title: Effect of Oxytocin Massage and Music on Breastfeeding: Randomized Controlled Trial
Brief Title: Effect of Oxytocin Massage and Music on Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elham Sadeghi, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IstUC
Record Dates: First submitted 2021-09-13; First posted 2021-09-28 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Oxytocin; Massage; Music; Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin massage (Active Comparator)
  Interventions: Other: Oxytocin massage AND music therapy
- music therapy (Active Comparator)
  Interventions: Other: Oxytocin massage AND music therapy
- control group (No Intervention)

INTERVENTIONS:
Other: Oxytocin massage AND music therapy — Oxytocin massage: It is a massage that will accelerate the work of the parasympathetic nerves in order to transmit the oxytocin production stimulus to the posterior lobe of the brain. Massage the scapula from the cervical 7th to the 5th-6th spine, spinal (vertebral), 1-2 cm around the spine, both thumbs up and then 2-3 times down, in a small circular clockwise, downward and upward movements. It is a form of massage by pressing hard.
  Music intervention: In order to decide on the type of music to be played to the mothers during breastfeeding, three samples (Pentatonic, Büzürk makam and classical music) selected by the researcher will be asked to the postpartum mother, and the music preferred by the mothers will be determined. It will be ensured that mothers listen to the music determined 5 minutes before the breastfeeding session for 7 days and continue breastfeeding while the same music is playing.
  Arms: Oxytocin massage; music therapy

SUMMARY:
The aim of this study is to examine the effect of oxytocin massage and music performed immediately after birth on breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* mothers who are 20 years or older,
* Primiparous delivery,
* Single fetus pregnancy,
* Born at term (38-42 weeks of gestation),
* Your baby's Apgar score is at least 8 points in the 5th minute,
* Being literate,
* Interviewed on the first day after birth,
* Does not have a problem that prevents breastfeeding,
* No complications during and after birth,
* Staying in the same room with her baby after birth,
* There is no health problem that may affect the baby's suckling,
* Those who become pregnant by normal means (without IVF, IVF, etc.),
* Babies with a birth weight of more than 2500,
* Mothers without chronic disease,
* Non-smoking mothers,
* Mothers who do not give formula to their babies

Exclusion Criteria:

* The mother/baby has a serious health problem that prevents breastfeeding,
* Absence from education for at least two sessions,
* Women with a known disease (HIV, hepatitis B, hepatitis C, etc.) known to be transmitted through breast milk will be excluded from the study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Diagnostic and Evaluation Scale | 1 month
  LATCH is a breastfeeding charting system that provides a systematic method for gathering information about individual breastfeeding sessions. The system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding. Each letter of the acronym LATCH denotes an area of assessment. "L" is for how well the infant latches onto the breast. "A" is for the amount of audible swallowing noted. "T" is for the mother's nipple type. "C" is for the mother's level of comfort. "H" is for the amount of help the mother needs to hold her infant to the breast. The minimum point is 0 and maximum point is 10. The highest 10 points to be obtained from the scale are taken, and a high score indicates good breastfeeding success.
Breastfeeding Self-Efficacy Scale short form | 1 month
  The questionnaire is a 14-item self-administered instrument derived from the original 33-items, that measures breastfeeding confidence. All items are preceded on a 5-point Likert scale, ranging from 1 to 5. Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy.
Infant Nutrition Attitude Scale | 1 month
  The scale is composed of 17 items with a 5-point Likert scale ranging from 1 to 5. The total IIFAS score can range from 17 to 85 with higher scores reflecting positive attitude towards breastfeeding. Total IIFAS scores can be further categorized into groups: 1) positive to breastfeeding (IIFAS score 70-85), 2) neutral (IIFAS score 49-69), and 3) positive to formula feeding (IIFAS score 17-48).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Other, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No